CLINICAL TRIAL: NCT03671577
Title: Building Closer Friendships in Social Anxiety Disorder: A Preliminary Test
Brief Title: Building Closer Friendships in Social Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Jesse Cougle, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018.23774
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Social Anxiety

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into active treatment or waitlist control.
Who Masked: Outcomes Assessor
Masking Description: Participants will be randomized into active treatment or waitlist control, so they will be aware of the condition they are in.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Experimental): four week computerized intervention designed to reduce fear of intimacy
  Interventions: Behavioral: Building Closer Friendships
- Wait List Control (No Intervention): Participants will continue as usual and will be given the option to receive the active treatment after completion of the study

INTERVENTIONS:
Behavioral: Building Closer Friendships — Intervention designed to build social support and reduce loneliness by giving participants skills to strengthen their relationships
  Arms: Active Treatment

SUMMARY:
This study assesses whether a 4-week computerized intervention can be used to decrease fear of intimacy, and loneliness and improve perceived social support in people with Social Anxiety Disorder.

DETAILED DESCRIPTION:
This study hopes to assess whether a month long computerized intervention aimed at giving people skills to form closer friendships. Participants will be randomized into an active treatment condition or a wait list control. We hypothesize that 1) participants in the treatment condition will have lower fear of intimacy at post treatment than those in the waitlist condition 2) participants in the treatment condition will have lower levels of loneliness than those in the waitlist condition 3) participants in the treatment condition will have higher perceived social support than those in the waitlist condition.

ELIGIBILITY:
Inclusion Criteria:

* Social Anxiety Disorder Diagnosed by the Mini International Neuropsychiatric Interview
* Social Phobia Inventory Score >19
* Stable psychotropic medication for the past month and kept stable for duration of study

Exclusion Criteria:

* Currently participating in therapy
* Current Substance Dependence
* Bipolar Disorder or psychotic illness
* Current suicidality (imminent risk)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Multidimensional Scale of Perceived Social Support | Change in Perceived Social Support from baseline to post treatment (4weeks) and one month follow up (8 weeks)
  Self-report scale that measures perceived levels of social support. Scores range from 12 to 84 with higher scores indicating higher levels of perceived social support. The three subscales (friends, family and significant other) all have a range of 4 to 28 with higher scores indicating higher levels of perceived social support.
Fear of Intimacy Scale-friend version | Change in fear of intimacy from baseline to post treatment (4weeks) and one month follow up (8 weeks)
  self report scale measuring fear of intimacy in friendships. Scores range from 26 to 130 with higher scores indicating a higher level of fear of intimacy.

SECONDARY OUTCOMES:
UCLA Loneliness Scale | Change in loneliness from baseline to post treatment (4weeks) and one month follow up (8 weeks)
  A 20 item Self report scale measuring loneliness. Scales range from 0 to 60 with higher scores indicating a higher level of loneliness.
Social Phobia inventory | Change in social anxiety symptoms from baseline to post treatment (4 weeks) and one month follow up (8 weeks)
  Self-report scale that measures Social anxiety symptoms. Scores range from 0 to 68 with higher scores indicating higher levels of social anxiety symptoms.
State-Trait Inventory for Cognitive and Somatic Anxiety-Trait Version (STICSA-T) | Change in overall anxiety symptoms from baseline to post treatment (4 weeks) and one month follow up (8 weeks)
  Self-report measure used to assess overall anxiety symptoms. Scores range from 21 to 84 with higher scores indicating higher levels of overall anxiety.
Center for Epidemiological Studies Depression Scale (CES-D) | Change in depression symptoms from baseline to post treatment (4 weeks) and one month follow up (8 weeks)
  Self-report measure used to assess depressive symptoms. Total scores range from 0 to 60 with higher scores indicating a higher level of depressive symptoms.
Interpersonal Needs Questionnaire (INQ) | Change in suicide vulnerability from baseline to post treatment (4 weeks) and one month follow up (8 weeks)
  Self report measure of suicide vulnerability. Total scores range from 15 to 105, with higher scores indicating a higher vulnerability for suicide.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States